CLINICAL TRIAL: NCT03462862
Title: Evaluation of Candida Albicans Growth on Bre.Flex Versus PEEK ( Polyether Ether Ketone ) Denture Base in Bilateral Maxillary Bounded Partial Denture (Randomized Clinical Trial)
Brief Title: Evaluation of Candida Albicans Growth on BreFlex Versus PEEK Denture Base in Maxillary Bounded Partial Denture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Sammy Mansour, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Peek vs Breflex
Record Dates: First submitted 2018-02-22; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Candida Albicans Infection
Keywords: PEEK; Breflex
MeSH Terms: interventions — polyetheretherketone

STUDY DESIGN:
Intervention Model Description: 2 parallel groups one group will receive RPD with PEEK denture base and the other will get Bre Flex denture base material
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): patients will receive partial denture constructed from PEEK material
  Interventions: Other: PEEK
- Group 2 (Active Comparator): patients will receive partial denture constructed from breflex material
  Interventions: Other: Bre-Flex

INTERVENTIONS:
Other: PEEK — PEEK has been successfully used over the last years in the medical ﬁeld, and orthopedics, speciﬁcally. which presents high bio compatibility, good mechanical properties, high temperature resistance, and chemical stability due to a 4 GPa modulus of elasticity, it is as elastic as bone and can reduce stresses transferred to the abutment teeth.Additional advantages of this polymer material are elimination of allergic reactions and metallic taste, high polishing qualities, low plaque afﬁnity, and good wear resistance, it has only recently been used in dentistry.
  Arms: Group 1
Other: Bre-Flex — In the recent time thermoplastic materials become quite popular in clinical practice such as nylon and acetal resins. since the 1950, poly-amide resin (nylons) provide improved esthetics and reduction of rotational forces on the abutment teeth due to their low elastic modulus(3).
  The major disadvantage of a nylon removable denture is the inability for a reline procedure and the lack of occlusal rests as well as rigid frameworks, that could lead to occlusal instability and sinking, especially in Kennedy class I and II cases. On the other hand, acetal resins present adequate mechanical strength to form a frame-work more rigid than nylon with retentive clasps, connectors, and supportive elements; however, the acetal resin material lacks natural translucency and vitality.
  Arms: Group 2

SUMMARY:
This study evaluate Candida Albicans growth on Bre-Flex versus PEEK denture base in Bilateral Maxillary bounded partial denture , half of patients will receive a framework with breflex denture base and the other half will receive a framework with PEEK denture base then evaluate the Candida growth

DETAILED DESCRIPTION:
Peek and Bre.flex are both new material that introduced to the market recently with great benefits like aesthetics and bio-compatibility but which material has less candida growth ? Bre.flex is a nylon-based thermoplastic material, composed of nylon polyamide 12 (polyamide).Nylon exhibits high physical strength, heat resistance and chemical resistance. It can be easily modified to increase stiffness and wear resistance. Nylon resin can be semi-translucent and provides excellent esthetics but it is a little more difficult to adjust and polish.

Despite of its highly esthetics features, Nylon still suffers from surface roughness that increase the colonization for candida but less than heat cured acrylic Recently, PEEK is introduced as a removable prosthesis material due to its high mechanical and biological properties but further clinical studies or systematic reviews focusing on the use of PEEK dentures are needed.

The patient will be treated in visits designated as follows:

Visit 1: Preoperative records, clinical, radiographic examination (panoramic and periapical x-rays for evaluation the crown-root ratio, the apical condition of the abutment and their alveolar bone support of abutment) and primary impression will be performed with irreversible hydro-colloid impression material (alginate), The impressions will be poured with type IV dental stone to obtain diagnostic casts.

Visit 2: Maxillary Face-bow will be recorded. The diagnostic casts will be mounted on semi adjustable articulator in centric occluding relation to evaluate the inter arch distance and occlusal plane.

Visit 3: primary surveying is performed. Special trays will be constructed and Mouth preparation will be performed by preparing guiding planes and rests seats on the abutments. Final impression will be taken by elastomeric impression material. The impression will be poured into type IV dental stone in order to obtain master cast. The master cast will be surveyed. The proposed design will be as follows: framework for edentulous areas on both sides connected with palatal strap. Aker's clasp on all abutments with buccal retention.

Visit 4: the metal framework is tried into the patient's mouth. Jaw relation is recorded.

Visit 5: The framework will be tried in with acrylic teeth in patient's mouth. Visit 6: the denture base of the partial denture will be processed incorporation with the metal framework into the two different materials to be evaluated. The first group will receive the partial denture in which the metal framework incorporated with the denture base fabricated from PEEK material. The second group will receive the partial denture in which the metal framework incorporated with the denture base material fabricated from BRE-FLEX.

Visit7, 8, 9: clinical measurement will be performed for one month in three visits.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have Kennedy class III modification I upper partially edentulous ridges.
* The remaining teeth have good periodontal condition, with no signs of attrition or gingival recession.
* Male or female patient with age range (30-55) and in good medical condition
* All patients have skeletal Angle's class I maxillo-mandibular relationship and have sufficient interarch distance.
* Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
* Free from any tempo-mandibular joint disorder.
* The patients have good oral hygiene and low caries index.

Exclusion Criteria:

* Patients having abnormal habits as bruxism or clenching
* Patients having hormonal disorders as diabetes, thyroid or parathyroid hormonal diseases were not included.
* Teeth with compromised bone support.
* Patient with xerostomia or excessive salivation.
* Patient with abnormal tongue behavior and/or size.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-06-28 (Estimated); Primary Completion 2018-07-22 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
Candida Albicans growth | one month
  after insertion of the denture we will measure the Candida count using Light Microscope and record the CFU/ML (colony-forming units per milliliter) unit

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Abbas, MD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Freitas Fernandes FS, Pereira-Cenci T, da Silva WJ, Filho AP, Straioto FG, Del Bel Cury AA. Efficacy of denture cleansers on Candida spp. biofilm formed on polyamide and polymethyl methacrylate resins. J Prosthet Dent. 2011 Jan;105(1):51-8. doi: 10.1016/S0022-3913(10)60192-8. PMID 21194588
- [Background] Guiotti AM, Goiato MC, Dos Santos DM, Vechiato-Filho AJ, Cunha BG, Paulini MB, Moreno A, de Almeida MT. Comparison of conventional and plant-extract disinfectant solutions on the hardness and color stability of a maxillofacial elastomer after artificial aging. J Prosthet Dent. 2016 Apr;115(4):501-8. doi: 10.1016/j.prosdent.2015.09.009. Epub 2015 Nov 19. PMID 26602149
- [Background] Parvizi A, Lindquist T, Schneider R, Williamson D, Boyer D, Dawson DV. Comparison of the dimensional accuracy of injection-molded denture base materials to that of conventional pressure-pack acrylic resin. J Prosthodont. 2004 Jun;13(2):83-9. doi: 10.1111/j.1532-849X.2004.04014.x. PMID 15210003
- [Background] Zoidis P, Papathanasiou I, Polyzois G. The Use of a Modified Poly-Ether-Ether-Ketone (PEEK) as an Alternative Framework Material for Removable Dental Prostheses. A Clinical Report. J Prosthodont. 2016 Oct;25(7):580-584. doi: 10.1111/jopr.12325. Epub 2015 Jul 27. PMID 26216668
- [Background] Pires FR, Santos EB, Bonan PR, De Almeida OP, Lopes MA. Denture stomatitis and salivary Candida in Brazilian edentulous patients. J Oral Rehabil. 2002 Nov;29(11):1115-9. doi: 10.1046/j.1365-2842.2002.00947.x. PMID 12453267